CLINICAL TRIAL: NCT04777656
Title: Randomized Trial for Unstable Pediatric Crohn's Disease Patients Comparing the Use of Crohn's Disease Exclusion Diet (CDED) on Top of Standard Therapy Versus Standard Therapy Alone.
Brief Title: Use of Crohn's Disease Exclusion Diet on Top of Standard Therapy Versus Standard Therapy Alone in Unstable Pediatric Crohn's Disease Patients.
Acronym: ASCENSION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other); MICALIS Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200010; 2020-A02569-30 (Other: ID-RCB)
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Recurrent inflammatory disorder; Immunomodulators; Biologics; Exclusive Enteral Nutrition; Crohn's disease exclusion diet (CDED); Modulen™IBD®
MeSH Terms: conditions — Crohn Disease | interventions — Maintenance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CDED/Modulen™IBD® (Experimental): Strategy combining CD exclusion diet plus Modulen™IBD® on top of ongoing maintenance therapy.
  Interventions: Dietary Supplement: Phase1 : CDED/Modulen™IBD® + Maintenance therapy; Dietary Supplement: Phase2 and 3 :
- Unrestricted food access (Active Comparator): Stop CDED and Modulen™IBD®, but continue maintenance therapy with unrestricted food access.
  Interventions: Dietary Supplement: Phase1 : CDED/Modulen™IBD® + Maintenance therapy
- Not randomized (Other): Patient not in remission at M2 or refusing randomisation
  Interventions: Dietary Supplement: Phase1 : CDED/Modulen™IBD® + Maintenance therapy

INTERVENTIONS:
Dietary Supplement: Phase1 : CDED/Modulen™IBD® + Maintenance therapy — from D0 until M2: Phase 1 (2 months run-in phase with CDED protocol + maintenance therapy, with the exception of corticosteroid that have to be tapered and stopped until M2.)
Dietary Supplement: Phase2 and 3 : — from M2 until M4 CDED phase 2 (introduction of a selected number of additional food). From M4 until end of the study CDED phase 3 (enlargement of number of additional foods and allowance of some initially excluded foods).
  Other Names: CDED/Modulen™IBD® + Maintenance therapy
  Arms: CDED/Modulen™IBD®

SUMMARY:
This research is a multicenter French randomized and single blinded phase III clinical trial evaluating two treatment strategies among Crohn's disease (CD) patients. The main objective is to assess if the addition of Crohn's Disease Exclusion Diet (CDED) to ongoing standard medication is superior to reduce the rate of relapses over 12 months compared to standard medication alone in children/adolescents with unstable CD responding with remission after a 2-months course of CDED

DETAILED DESCRIPTION:
Crohn's disease is a recurrent inflammatory disorder. Current treatment strategies aim reducing intestinal (and systemic) inflammation based on the use of Immunomodulators (IM) and biologics (B). However, some patients, particularly in the pediatric age group do not respond with remission to standard therapy and approximately 30% of patients lose response to efficient therapy. There is a clear unmet need for new treatment strategies. In addition, patients and families have a high degree of reluctance to use IM/B as life-long medication, particularly due to potential side effects including cancer, lymphomas, serious infections or drug-related immune diseases. This is of particular importance for children/adolescents with CD, potentially exposed over many decades to various IM/B. Experimental and epidemiological data indicate that the western life style and particularly modern food play a key role in the development of CD, probably via alteration of the intestinal barrier function and/or enforcing the intestinal dysbiosis. Based on these data and the observation that exclusive enteral nutrition is highly efficacious in inducing remission in active CD, nutritional therapies are more and more in the focus for the development of new treatment approaches.

The main objective is to assess if the addition of CDED to ongoing standard medication is superior to reduce the rate of relapses over 12 months compared to standard medication alone in children/adolescents with unstable CD responding with remission after a 2-months course of CDED.

To achieve this objective, eligible patients with active CD will participate to this study for a 13 months period. After a screening period, the patients will have a 2 months run-in phase where they will follow the CDED protocol, but continue their maintenance therapy, with the exception of corticosteroid that have to be tapered and stopped at the end of the 2 months.

Then, the patients responding to CDED during run-in will be randomized at M2 to one of the two treatment arms (CDED/Modulen™IBD® or Unrestricted food access) and will have 4 follow-up visits (M4, M6, M9 and M12)

ELIGIBILITY:
Inclusion Criteria:

* Child/Adolescent aged 6-17 years with a confirmed diagnosis of CD (for at least 3 months) with an active disease (defined as: wPCDAI >12.5 or CRP > 2 times upper limit or calprotectin levels >250µg/g if available) despite anti-inflammatory (5-ASA and derivates), corticosteroids, immunomodulator (thiopurines or methotrexate) and/or biologic therapy (anti-TNF, anti-integrin anti-IL23 antibodies)
* For girls of childbearing age: a negative pregnancy test, and use of an effective method of contraception (abstinence, oral contraceptives, intra-uterine device, diaphragm with spermicide and condom)
* Patient willing to comply with daily intake of an exclusion diet
* Informed and signed consent of parents
* Patient affiliated to social security (or health insurance)

Exclusion Criteria:

* Active perianal fistulizing disease
* Internal fistula or evidence of un-drained and un-controlled abscess/phlegmon
* Patient who require CD-related surgical therapy
* Patient with known allergy to cow milk's proteins
* Patient incapable to follow CDED for a prolonged period
* Pregnancy, breastfeeding
* Patient already included in an interventional study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Relapse from randomization until M12 | 12 months
  Relapse is defined as weighted Paediatric Crohn's disease activity index (wPCDAI) >40 points and/or CRP >2 times over upper limit (in the absence of any obvious infections sign) or if at two consecutive visits (within 2-8 weeks) the wPCDAI is >12,5 but less 40 and/or CRP >1,5 but less 2 times over upper limit (in the absence of any obvious infections sign) or if the patient required additional CD-specific medication/surgery in the interval.

SECONDARY OUTCOMES:
Change of wPCDAI from baseline to M2 | 2 months
Change of fecal calprotectin values from baseline to M2 | 2 months
Clinical remission at M2 | 2 months
  Defined as wPCDAI ≤12.5 and normal CRP (≤1.5 fold upper normal range)
Deep remission at M2 | 2 months
  Defined as wPCDAI ≤12.5 and normal CRP within normal lab range) and normal fecal calprotectin ((<250µg/g)
Physician global assessment (PGA) from baseline to M2 | 2 months
  Crohn's Disease activity assessed as remission - weak - moderate - severe
Mucosal healing at M2 | 2 months
  absence of any ulcerations (including aphthae)
Endoscopic response at M2 | 2 months
  Decrease of Crohn's Disease Endoscopic Index Score (CDEIS) ≥ 50% from baseline
Change of MRI from baseline to M2 | 2 months
  Simplified Magnetic Resonance Index of Activity (MARIA) for Crohn's Disease score from baseline to M2
CDED tolerance rate at M2 | 2 months
  serious and non serious adverse events
CDED compliance rate at M2 | 2 months
Change of intestinal microbiome composition from baseline to M2 | 2 months
Clinical remission | At 4 months, 6 months, 9 months and 12 months
  Defined as wPCDAI ≤12.5 and normal CRP (≤1.5 fold upper normal range)
Deep remission | At 4 months, 6 months, 9 months and 12 months
  Defined as wPCDAI ≤12.5 and normal CRP (within normal lab range) and normal fecal calprotectin (<250µg/g)
Relapse | At 4 months, 6 months, 9 months and 12 months
  Defined as wPCDAI >40 points and/or CRP >2 times over upper limit (in the absence of any obvious infections sign) or if at two consecutive visits (within 2-8 weeks) the wPCDAI is >12,5 but less 40 and/or CRP >1,5 but less 2 times over upper limit (in the absence of any obvious infections sign) or if the patient required additional CD-specific medication/surgery in the interval
Physician global assessment (PGA) | At 4 months, 6 months, 9 months and 12 months
  Crohn's Disease activity assessed as remission - weak - moderate - severe
Mucosal Healing at M12 | 12 months
  Absence of any ulcerations (including aphthae)
Endoscopic response at M12 | 12 months
  Decrease of Crohn's Disease Endoscopic Index Score (CDEIS) ≥ 50% from baseline
Change of MRI from M2 to M12 | 12 months
  Simplified Magnetic Resonance Index of Activity (MARIA) for Crohn's Disease score from M2 to M12
CDED tolerance rate at M12 | 12 months
  Serious and non serious adverse events
CDED compliance rate at M12 | 12 months
Change of Intestinal microbiome composition | At 4 months, 6 months, 9 months, 12 months
Change of quality of life IMPACT-3 from inclusion until 12 months | At baseline, 2 months, 4 months, 6 months, 9 months, 12 months
  IMPACT-3 questionnaire of 35 closed questions - scale ranging from 1 to 5 for all answers - higher score suggesting better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Franck Ruemmele, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hôpital Femme mère enfant, CHU Lyon - Service Hépato-gastroentérologie et Nutrition pédiatrique, Bron
  - CHU Caen Normandie - Service de Gastroentérologie pédiatrique, Caen
  - Hôpital de la Timone, AP-HM - Service de Gastroentérologie pédiatrique, Marseille
  - Hôpital Necker-Enfants malades - Service de Gastroentérologie pédiatrique, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruemmele FM, Veres G, Kolho KL, Griffiths A, Levine A, Escher JC, Amil Dias J, Barabino A, Braegger CP, Bronsky J, Buderus S, Martin-de-Carpi J, De Ridder L, Fagerberg UL, Hugot JP, Kierkus J, Kolacek S, Koletzko S, Lionetti P, Miele E, Navas Lopez VM, Paerregaard A, Russell RK, Serban DE, Shaoul R, Van Rheenen P, Veereman G, Weiss B, Wilson D, Dignass A, Eliakim A, Winter H, Turner D; European Crohn's and Colitis Organisation; European Society of Pediatric Gastroenterology, Hepatology and Nutrition. Consensus guidelines of ECCO/ESPGHAN on the medical management of pediatric Crohn's disease. J Crohns Colitis. 2014 Oct;8(10):1179-207. doi: 10.1016/j.crohns.2014.04.005. Epub 2014 Jun 6. PMID 24909831
- [Background] Wynands J, Belbouab R, Candon S, Talbotec C, Mougenot JF, Chatenoud L, Schmitz J, Cezard JP, Goulet O, Hugot JP, Ruemmele FM. 12-month follow-up after successful infliximab therapy in pediatric crohn disease. J Pediatr Gastroenterol Nutr. 2008 Mar;46(3):293-8. doi: 10.1097/MPG.0b013e31815604cd. PMID 18376247
- [Background] Pigneur B, Lepage P, Mondot S, Schmitz J, Goulet O, Dore J, Ruemmele FM. Mucosal Healing and Bacterial Composition in Response to Enteral Nutrition Vs Steroid-based Induction Therapy-A Randomised Prospective Clinical Trial in Children With Crohn's Disease. J Crohns Colitis. 2019 Jul 25;13(7):846-855. doi: 10.1093/ecco-jcc/jjy207. PMID 30541015
- [Background] Levine A, Wine E, Assa A, Sigall Boneh R, Shaoul R, Kori M, Cohen S, Peleg S, Shamaly H, On A, Millman P, Abramas L, Ziv-Baran T, Grant S, Abitbol G, Dunn KA, Bielawski JP, Van Limbergen J. Crohn's Disease Exclusion Diet Plus Partial Enteral Nutrition Induces Sustained Remission in a Randomized Controlled Trial. Gastroenterology. 2019 Aug;157(2):440-450.e8. doi: 10.1053/j.gastro.2019.04.021. Epub 2019 Jun 4. PMID 31170412
- [Background] Levine A, Sigall Boneh R, Wine E. Evolving role of diet in the pathogenesis and treatment of inflammatory bowel diseases. Gut. 2018 Sep;67(9):1726-1738. doi: 10.1136/gutjnl-2017-315866. Epub 2018 May 18. PMID 29777041